CLINICAL TRIAL: NCT02487589
Title: Feasibility and Cost-effectiveness of a Multidisciplinary Home-telehealth Intervention Programme to Reduce Falls Among Elderly Discharged From Hospital: a Randomized Controlled Trial
Brief Title: Falls in Elderly and Telehealth: a Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Alessandro Giordano, Medical Doctor, Fondazione Salvatore Maugeri
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GR-2010-2310662
Record Dates: First submitted 2015-06-18; First posted 2015-07-01 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Diseases
Keywords: Falls; Elderly; e-Health; Telemedicine
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): In Italy, medical risks and patients risk behaviour are not systematically registered and addressed by hospital physicians, specialists and general practitioners (GPs).
  Patients allocated in control group will receive by the hospital staff tailored recommendations based on their own risk profile. The same information will be sent to their GPs. No restrictions on co-interventions will be placed.
- Treated group (Experimental): Telephone support, telemonitoring and tele-exercise
  Interventions: Other: Telephone support, telemonitoring and tele-exercise

INTERVENTIONS:
Other: Telephone support, telemonitoring and tele-exercise — The care model will provide 24/24 h assistance for six months and include:
  Telephone Support: a nurse-tutor (NT) will follow-up the enrolled patients weekly mainly through scheduled appointments. NTs duties will be: 1 education (patients and family ' s health education on how to prevent falls, verification of the adherence to the pharmacological therapy, teaching on how to recognize problems that can conduct to falls) and 2. management. Occasional appointments will be required by patients on duty and managed by a nurse .
  Telemonitoring: all patients will send proper biological traces and data will be registered on a personal health record.
  Tele-exercise: Home exercises sessions will be provided by a DVD and monitored through a videoconference by a physiotherapist.
  Arms: Treated group

SUMMARY:
Fall incidents are the third cause of chronic disablement in elderly according to the World Health Organization (WHO). Recent meta-analyses shows that a multifactorial falls risk assessment and management programs are effective in all older population studied. However, the application of these programs may not be the same in all National health care setting and, consequently, needs to be evacuated by cost-effectiveness studies before to plan this intervention in regular care. In Italy structured collaboration between hospital staff and primary care is generally lacking and the role of Information and Communication Technologies (ICT) in a fall prevention program at home has never been explored.

This is a two-group randomized controlled trial aiming to evaluate the effect of a home-based intervention program, delivered by a multidisciplinary health team, in preventing falls in elderly. The home tele-management program, previously adopted in our Institute for chronic patients, will be proposed to elderly people affected by chronic diseases at high risk of falling at time of hospital discharge. The program will involve the hospital staff and will be managed thanks to the collaboration between hospital and primary care setting. Patients will be followed at home for 6 months after hospital discharge. A nurse-tutor will be the case manager and telephone support, telemonitoring and tele-exercise will characterize the intervention program. People in the control group will receive the usual care. The main outcome measure of the study will be the percentage of patients sustaining a fall during the 6-months follow-up period. An economic evaluation will be performed from a societal perspective and will involve calculating cost-effectiveness and cost utility ratios.

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the effects of a home-based intervention program delivered by a multidisciplinary team through available ICT on recurrent falls in elderly discharged from hospital. This objective results in the following research questions:

Is the program more effective than usual care in preventing new falls after hospital discharge?

Is the program cost-effective compared to usual care when assessed from a community perspective?

Besides the effect and economic evaluations, a process evaluation will be carried out to assess the feasibility and the applicability of the program for those receiving and implementing the intervention.

The investigators expect that an intervention program can be effective to reduce falls in elderly patients discharged from hospital. The feasibility of the program for the participants and the cost-effectiveness analysis will confirm whether or a larger national trial is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and over
* Patients with a high risk profile (at least one fall event in the last 12 months, Berg scale score ≤ 45 and at least one fall event during in-hospital stay) of recurrent falling
* Patients discharged from the Institute of Fondazione Salvatore Maugeri, IRCCS after a period of rehabilitation and living independently

Exclusion Criteria:

* Patients' inability to sign the informed consent
* Patients living in a nursing home
* Patients permanently bedridden or fully dependent on a wheelchair
* Patients with cancer
* Patients with Mini Mental Examination State (MMSE) < 18
* Patients with MMSE < 24 lacking of caregiver at home
* Patients with neurological impairment (i.e. aphasia and neglect)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 280 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Falls events | 6-months
  The percentage of patients sustaining a fall

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Giordano, MD, Principal Investigator — Fondazione Salvatore Maugeri
Locations (1):
- Fondazione Salvatore Maugeri, IRCCS, Lumezzane, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giordano A, Bonometti GP, Vanoglio F, Paneroni M, Bernocchi P, Comini L, Giordano A. Feasibility and cost-effectiveness of a multidisciplinary home-telehealth intervention programme to reduce falls among elderly discharged from hospital: study protocol for a randomized controlled trial. BMC Geriatr. 2016 Dec 7;16(1):209. doi: 10.1186/s12877-016-0378-z. PMID 27923343